CLINICAL TRIAL: NCT05836142
Title: Stabilometry and Plantar Pressures Changes After Progressive Pressure Release in Flexor Digitoum Brevis in Latent Trigger Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayuben Private Clinic (Other)
Responsible Party: Principal Investigator, EVA MARIA MARTÍNEZ JIMENEZ, Head of Podiatry, Principal Investigator, and Physiotherapist, Mayuben Private Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1912202200923
Record Dates: First submitted 2023-04-18; First posted 2023-05-01 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Bilateral Latent Myofascial Trigger Points of Flexor Digitorum Brevis
Keywords: Foot; Stabilometry; Platform; therapeutics; trigger point

STUDY DESIGN:
Intervention Model Description: Pretest posttest of bilateral Flexor digitorum Brevis progressive pressure release intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: progressive pressure release (Experimental): Bilateral progressive pressure release in latent trigger points of the Flexor digitorum Brevis Muscle
  Interventions: Procedure: progressive pressure release

INTERVENTIONS:
Procedure: progressive pressure release — Bilateral progressive pressure release in latent trigger points of the Flexor digitorum Brevis Muscle

SUMMARY:
The aim of this clinical trial is to check the effects of progressive pressure release in the Flexor digitorum Brevis

DETAILED DESCRIPTION:
Eighteen subjects with bilatereal lantent myofascial trigger points wil be recruited for a pre- test post-test study. Participants will be from 18 to 40 years old, not obese. Participants will be measured before and after bilateral dry needling in Flexor digitorum Brevis. The investigators will measure stabilometry variables and static footprint. The footprint variables will be divided in bilateral rear foot, bilateral midfoot, bilateral fore foot.

Stabilometry will be measured by displacement of the center of pressures in X and Y with eyes open and closed , center of pressure (COP) with eyes open and closed, COP area with eyes open and closed, COP antero-posterior (a-p) and medio-lateral (m-lat) directions with eyes open and closed, and COP speed. Two trials will be recorded for each condition and the order of the conditions will be randomized across subjects, eyes open and eyes closed. Foot plantar pressure and surface area of two static footprints will be measured during bipedal standing. Static plantar pressure will be evaluated by means of maximum pressure, medium pressure and surface area of each aspect of the foot (rearfoot, midfoot, and fore foot).

ELIGIBILITY:
Inclusion Criteria:

* Asyntomatic subjects with flat foot

Exclusion Criteria:

* Previous lower extremities surgery. History of lower extremities injury with residual symptoms (pain, "giving-away" sensations) within the last year.

Leg-length discrepancy more than 1 cm Balance deficits (determined by oral questionnaire regarding falls)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-05-27 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
Static footprint | Through study completion, an average of 3 days
  Static footprint will measure plantar presures and surface area of rear food, midfoot and fore foot. Subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. During all the examinations, the upper limbs were placed in a relaxed position along the body. The subjects were instructed to stand as still as possible for 30 s, with their eyes open, while concentrating on a point at eye level 2-m away or with their eyes open.
Stabilometry variable x displacement open eyes before progressive pressure release | Through study completion, an average of 3 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of pressures in X (in milimeters) with open eyes.
Stabilometry variable y displacement open eyes before progressive pressure release | Through study completion, an average of 3 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of pressures in Y (in milimeters) with open eyes.
Stabilometry variable center of pressure area open eyes before progressive pressure release | Through study completion, an average of 3 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of Pressure (COP) area (in milimeters²) with eyes open.
Stabilometry variable center of pressure speed displacement of the anteroposterior(a-p) direction open eyes before progressive pressure release | Through study completion, an average of 3 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure center of pressure speed displacement of the anteroposterior(a-p) direction (in milimeters/second).
Stabilometry variable center of pressure speed displacement of the latero-lateral(lat-lat) direction open eyes before progressive pressure release | Through study completion, an average of 3 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure center of pressure speed displacement of the latero-lateral(lat-lat) direction (in milimeters/second).
Stabilometry variable x displacement before progressive pressure release with closed eyes | Through study completion, an average of 3 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of pressures in X (in milimeters) with eyes closed.
Stabilometry variable y displacement before progressive pressure release with closed eyes | Through study completion, an average of 3 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of pressures in Y (in milimeters) with closed eyes.
Stabilometry variable center of pressure area before progressive pressure release with closed eyes | Through study completion, an average of 3 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of Pressure (COP) area (in milimeters²) with eyes closed.
Stabilometry variable center of pressure speed displacement of the anteroposterior(a-p) direction before progressive pressure release with closed eyes | Through study completion, an average of 3 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure center of pressure speed displacement of the anteroposterior(a-p) direction (in milimeters/second).
Stabilometry variable center of pressure speed displacement of the latero-lateral(lat-lat) direction before progressive pressure release with closed eyes | Through study completion, an average of 3 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure center of pressure speed displacement of the latero-lateral(lat-lat) direction (in milimeters/second).
Stabilometry variable x displacement open eyes after intervention | Through study completion, an average of 3 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of pressures in X (in milimeters) with open eyes.
Stabilometry variable y displacement open eyes after intervention | Through study completion, an average of 3 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of pressures in Y (in milimeters) with open eyes.
Stabilometry variable center of pressure area open eyes after intervention | Through study completion, an average of 3 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of Pressure (COP) area (in milimeters²) with eyes open.
Stabilometry variable center of pressure speed displacement of the anteroposterior(a-p) direction with open eyes after intervention | Through study completion, an average of 3 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure center of pressure speed displacement of the anteroposterior(a-p) direction (in milimeters/second).
Stabilometry variable center of pressure speed displacement of the latero-lateral(lat-lat) direction with open eyes after intervention | Through study completion, an average of 3 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure center of pressure speed displacement of the latero-lateral(lat-lat) direction (in milimeters/second).
Stabilometry variable x displacement with closed eyes after intervention | Through study completion, an average of 3 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of pressures in X (in milimeters) with eyes closed.
Stabilometry variable y displacement with closed eyes after intervention | Through study completion, an average of 3 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of pressures in Y (in milimeters) with closed eyes.
Stabilometry variable center of pressure area with closed eyes after intervention | Through study completion, an average of 3 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of Pressure (COP) area (in milimeters²) with eyes closed.
Stabilometry variable center of pressure speed displacement of the anteroposterior(a-p) direction with closed eyes after intervention | Through study completion, an average of 3 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure center of pressure speed displacement of the anteroposterior(a-p) direction (in milimeters/second).
Stabilometry variable center of pressure speed displacement of the latero-lateral(lat-lat) direction with closed eyes after intervention | Through study completion, an average of 3 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure center of pressure speed displacement of the latero-lateral(lat-lat) direction (in milimeters/second).

CONTACTS AND LOCATIONS:
Locations (1):
- Eva María Martínez-Jiménez In Mayuben CLinic, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No